CLINICAL TRIAL: NCT02227823
Title: Safety and Efficacy Study of Anti-cholinesterase Therapy on the Motor Functions in Patients With Spinal Muscular Atrophy Type 3.
Brief Title: Safety and Efficacy Study of Pyridostigmine on Patients With Spinal Muscular Atrophy Type 3
Acronym: EMOTAS
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Centre Hospitalier Régional de la Citadelle (Other)
Responsible Party: Principal Investigator, Dr. Stéphanie Delstanche, Neurologist, Centre Hospitalier Régional de la Citadelle
Allocation: Non-Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: 1376
Record Dates: First submitted 2014-08-20; First posted 2014-08-28 (Estimated); Last update posted 2023-10-11 (Actual); Status verified 2023-10

CONDITIONS: Spinal Muscular Atrophy Type 3
Keywords: spinal muscular atrophy type 3; electromyography; fatigability; decrement
MeSH Terms: conditions — Spinal Muscular Atrophies of Childhood | interventions — Pyridostigmine Bromide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- significant decrement (Experimental): Patients with significant decrement at electromyogram will be treated by pyridostigmine bromide 60mg 3 times a day for patients older than 18 and 1.5mg/kg 3 times a day for children less than 40kg
  Interventions: Drug: Pyridostigmine Bromide
- no decrement (No Intervention): Patient without significant decrement will not receive any treatment and will be the control group

INTERVENTIONS:
Drug: Pyridostigmine Bromide
  Other Names: Mestinon
  Arms: significant decrement

SUMMARY:
The purpose of this study is to evaluate safety and efficacy of anti-cholinesterase therapy on the motor function in SMA type 3 patients with impaired neuromuscular junction (NMJ).

DETAILED DESCRIPTION:
Spinal muscular atrophy (SMA) is the second neuromuscular disease meet in children. SMA is a genetically transmitted disease inducing muscular weakness predominating on shoulders and hips. Currently, there is no effective therapy to slow the progression of the disease. SMA is due to a neuron motor attempt of the spinal cord and recently it has been demonstrated a neuromuscular junction (NMJ) involvement, according to recent studies.

EMOTAS study aim to understand if NMJ abnormalities could have an impact on motor performance and fatigue in SMA type 3 ambulatory patients by electromyogram and to improve by non-invasive therapy quality of life of patients.

ELIGIBILITY:
Inclusion Criteria:

* Spinal muscular atrophy type 3, genetically confirmed

  * Age higher than 6 years old
  * Ambulatory patient
  * Informed consent signed
  * More than 100 meters of walking at 6-minute walk test at screening
  * Value at screening and baseline in a range of 20% of the highest value at 6-minute walk test

Exclusion Criteria:

* Patient who had surgical intervention or suffer from a recent traumatism (less than 6 months)

  * Associated pathology such as endocrinopathy, infectious disease, allergy, myopathy, chronic or acute inflammatory pathology, during 3 weeks preceding the inclusion.
  * Other therapeutics than food supplements or those frequently prescribed in spinal muscular atrophy or its complications
  * Non tolerance of electromyography
  * Limited collaboration due to trouble in information comprehension
  * Pathology inducing contra-indication for pyridostigmine treatment (allergy at molecule, asthma, Parkinson disease, mechanic obstruction of urinary or digestive tracts)

Min Age: 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2014-07; Primary Completion 2017-07 (Actual); Study Completion 2017-07 (Actual)

PRIMARY OUTCOMES:
Change from Baseline in the distance walked at 6-minute walk test at 6 months | 6 months

SECONDARY OUTCOMES:
Change from baseline of decrement at 6 months | 6 months
Change from baseline of MFM-D1 | 6 months
  Comparison of treated and control group values will be made
Change from baseline of Moviplate values at 6 months | 6 months
  Comparison between treated and control group value will be made
Change from baseline of the ratio at 6 minutes walk test at 6 months | 6 months
  It's the ratio between the number of meters during the last minute of the 6-minute walk test and the first minute of the 6-minute walk test.

CONTACTS AND LOCATIONS:
Overall Officials: Stephanie Delstanche, Principal Investigator — Centre de référence des maladies neuromusculaire de Liège
Locations (1):
- Centre de référence des maladies neuromusculaire, Centre Hospitalier Régional de la Citadelle, Liège, Belgium